CLINICAL TRIAL: NCT06206005
Title: Clinical and Radiographic Outcomes Around Four Mandibular Implant-retained Overdentures in Individuals With Type 2 Diabetes: A Long-term Retrospective Preliminary Study
Brief Title: Four Mandibular Implant-retained Overdentures in Individuals With Type 2 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Collaborators: Menoufia University (Other)
Responsible Party: Principal Investigator, Mohamed Elsawy, lecturer, Department of prosthodontics, principle investigator, Mansoura University
Other Study IDs: A03012023RP
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Bone Resorption
MeSH Terms: conditions — Bone Resorption | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group1 with Haemoglobin A1c ≤6.5%: This group represents a well-controlled type 2 Diabetics mellitus.
  Interventions: Other: Observational study
- Group 2 with Haemoglobin A1c >6.5%: This group represents a poorly controlled type 2 Diabetics mellitus.
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — evaluate implant survival, peri-implant outcome of 4 implant retained mandibular OVD after 10 years of function.

SUMMARY:
Studies clinically evaluate the long-term outcome of 4 implant attachment-retained mandibular OVDs among patients with high glycemic levels are lacking.

DETAILED DESCRIPTION:
Chronic hyperglycemia is considered as a typical risk-factor that causes soft tissue inflammation and bone loss around natural teeth and implants. One possible explanation for this mechanism is that chronic hyperglycemia has the propensity to increase the levels of accumulated glycation end products (AGEs) in the serum and oral tissues that accelerates the production of proinflammatory cytokines that induce bone destruction around natural teeth and implants. However, it is relevant to indicate that dental implants in chronic hyperglycemia under ideal glycemic conditions can successfully osseointegrate and show predictable outcomes over long durations in both diabetic and non-diabetic patients.

Studies clinically evaluate the long-term outcome of 4 implant attachment-retained mandibular OVDs among patients with high glycemic levels are lacking.

ELIGIBILITY:
Inclusion Criteria:

* Patients with edentulous maxilla and mandible for at least 12 months.
* Patients have problems with mandibular denture retention and stability.
* Patients with a mandibular bone height measured on a panoramic x-ray between 15 and 25 mm at the mandibular symphysis region.

Exclusion Criteria:

* Patients who did not receive implants at the department clinic.
* Patients with more or less than 4 implants in the mandible.
* Patients with well controlled diabetics.
* Patients with relative contraindications, such as a history of parafunctional habits, daily smokers of more than 10 cigarettes, or alcoholism.
* Patients who have previously received head and neck radiation therapy; furthermore, patients receiving intravenous bisphosphonates, chemotherapy, or psychological disorders could jeopardize their cooperation.

Ages: 55 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 20 participants at least.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-05-05 (Estimated); Study Completion 2024-08-05 (Estimated)

PRIMARY OUTCOMES:
Crestal bone loss around implants | This is a retrospective study, Measurement will be performed after implants being in service by 10 years
  amount of bone loss which appears on a periapical radiograph

SECONDARY OUTCOMES:
Probing depth | This is a retrospective study, Measurement will be performed after implants being in service by 10 years
  By using a plastic periodontal probe to measure the probing depth around the implants

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammed ELSawy, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No
The IPD is upon request from the corresponding author